CLINICAL TRIAL: NCT01249456
Title: An Observational, Multicenter Study on the Safety and Efficacy of Femara(Letrozole) as an Extended Adjuvant Treatment in Breast Cancer Patients Who Completed Adjuvant Tamoxifen or Toremifen Treatment
Brief Title: Safety and Efficacy Study of Femara(Letrozole) as an Extended Adjuvant Treatment in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CFEM345DKR04
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Letrozole
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Femara(Letrozole)

SUMMARY:
Title of study: An observational, multicenter study on the safety and efficacy of Femara® (Letrozole) as an extended adjuvant treatment in breast cancer patients who completed adjuvant Tamoxifen or Toremifen treatment

Objectives:

The major objective of the study is to assess safety and efficacy of Femara® in women who had undergone resection of a primary breast cancer and subsequently received prior adjuvant tamoxifen or toremifen therapy for 5 years in real-life condition.

The study aims at the following objectives:

1. To identify unknown adverse reactions, especially serious adverse reactions
2. To evaluate incidence and descriptions of adverse reactions under the routine drug use
3. To identify factors that may affect the safety of Femara®
4. To identify factors that may affect the efficacy of Femara®

Methodology: This will be an open-label, multi-center, single-arm, observational phase IV study.

Number of centers & patients: Approximately 610 (planned No. of patients for total study period) patients from 4 centers will be enrolled in this study.

Population: Postmenopausal early breast cancer patients who have finished adjuvant treatment with Tamoxifen or Toremifen for 5 years after curative surgery as "indications" described in local product labeling.

Investigational drug: Femara® will be administered orally as described in "dose & administration" of local product labeling up to 3 years.

Study duration: FPFV May. 2006, LPFV Dec. 2011. Study drug will be administered for up to 3 years with renewal of contract on yearly basis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent form
* Postmenopausal patients who had had a histologically or cytologically confirmed breast cancer removed at the time of diagnosis with no evidence of metastases and who had completed over 5 years of adjuvant therapy with tamoxifen or toremifen before entering the study
* Age ≥50 years with cessation of menses and Age <50 years Postmenopausal status defined by one of the following:

  * FSH level > 30-40 IU/L
  * cessation of menses over the past 1 year
  * are/become amenorrheic due to either chemotherapy or LHRH, are/become amenorrheic due to surgical ovarian ablation
* The tumor was to be ER and/or PgR-positive or the receptor status could have been unknown
* No evidence of recurrence of the disease at entry
* Patient must be accessible for follow-up

Exclusion Criteria:

* Those patients known to have had receptor-negative primary tumors
* Any concurrent malignancy
* Patients who previously received hormone replacement therapy (HRT) during 5 years of adjuvant therapy with tamoxifen or toremifen
* Patients who are currently receiving other aromatase inhibitors, or chemotherapy
* Patients who have serious cardiovascular or hepatic disease with significantly abnormal daily function and/or laboratory results
* Life expectancy < 12 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Postmenopausal early breast cancer patients who have finished adjuvant treatment with Tamoxifen or Toremifen for 5 years after curative surgery as "indications" described in local product labeling
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2006-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To identify unknown adverse reactions, especially serious adverse reactions | for 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea